CLINICAL TRIAL: NCT01794325
Title: Transradial and Transfemoral Approach by EXPERienced Operators in Daily rouTine (EXPERT): a Randomized, Non-inferiority Trial
Brief Title: Transradial and Transfemoral Coronary Angiography by EXPERienced operaTors
Acronym: EXPERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Hospital Ernesto Dornelles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP 4786/12
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Exposure to Ionizing Radiation; Coronary Heart Disease; Vascular Access Complication
Keywords: Occupational radiation exposure; Transradial approach; Transfemoral approach
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trans-radial access (Active Comparator): Coronary angiography performed through trans-radial access
  Interventions: Other: Trans-radial
- Trans-femoral access (Active Comparator): Coronary angiography performed through trans-femoral access
  Interventions: Other: Trans-femoral

INTERVENTIONS:
Other: Trans-radial — Coronary angiography performed through trans-radial access
  Arms: Trans-radial access
Other: Trans-femoral — Coronary angiography performed through trans-femoral access
  Arms: Trans-femoral access

SUMMARY:
Transradial approach (TRA) reduces vascular complications and access related-bleeding compared to transfemoral approach (TFA). However, this technique has been related to higher radiation exposure during coronary angiography and percutaneous coronary intervention. Previous studies have shown that TRA demands a long learning curve, and procedure success rate increases with operator's experience. Our hypothesis is that the higher radiation exposure during TRA is not a technique issue, but due to operator's expertise.

The aim of this study is to evaluate whether experienced operators with either TRA or TFA can perform diagnostic coronary angiography with similar radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a elective coronary angiography
* Eligible for either transfemoral or transradial approach
* Accept to sign the written consent form (WCF)

Exclusion Criteria:

* Refusal to sign the WCF
* End stage renal failure
* Urgency/Emergency procedure
* Contraindication to perform both coronary and left ventricle angiogram
* Necessity of another vascular angiogram during coronary angiography

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Patient radiation exposure (mGy) | during coronary angiography
  Patient radiation exposure (mGy)

SECONDARY OUTCOMES:
Physician radiation exposure (in uSv) | during coronary angiography
  Physician radiation exposure (in uSv)

OTHER OUTCOMES:
Major adverse cardiac events | 30 days
  Major adverse cardiac events (death, stroke and vascular complications)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano O Cardoso, MD, MSc, Study Chair — Instituto de Cardiologia do Rio Grande do Sul; Luis M Yordi, MD, Study Director — Hospital Ernesto Dornelles; Claudio V Moraes, MD, Principal Investigator — Insituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil